CLINICAL TRIAL: NCT06240078
Title: Impact of Chronic Obstructive Pulmonary Disease (COPD) on Sexual Health, Loneliness, and Well-being: A Cross-sectional Study of Prevalence and Associated Variables in Individuals With and Without COPD
Brief Title: Impact of COPD on Sexual Health, Loneliness, and Well-being
Status: Completed | Type: Observational
Sponsor: Vejle Hospital (Other)
Collaborators: Region of Southern Denmark (Other)
Responsible Party: Sponsor
Other Study IDs: COPD and sexual health
Record Dates: First submitted 2024-01-25; First posted 2024-02-02 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Sexual Health; Loneliness; Well-Being, Psychological
Keywords: COPD; sexual distress; sexual health; anxiety; depression; loneliness; chronic; associations
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Psychological Well-Being; Anxiety Disorders; Depression; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COPD group: COPD group: Participants with self-reported COPD (Group 1)
- Non-COPD group: Non-COPD group: Participants without self-reported COPD, but with other chronic diseases. A comparison group (Group 2)

SUMMARY:
Summary Person-centered care is a hot topic within healthcare, yet communication about patients' sexual health and intimacy issues remain too hot to handle within healthcare. Research indicates that sexual dysfunction and impaired sexual health are frequent among individuals with chronic obstructive pulmonary disease (COPD). Despite patients expecting healthcare professionals to address intimacy issues; these issues are often neglected, since the topic is a taboo.

This study aims to address a gap in observational research by investigating the physical, psychological and social aspects of sexual health in both men and women with and without COPD. The primary hypothesis of this survey-based cross-sectional study is that COPD negatively impacts sexual health, leading to increased loneliness, relationship dissatisfaction, anxiety and/or depression, along with decreased health-related quality of life and well-being in patients. The study seeks to identify associations between impaired sexual health and these factors.

By fostering a new understanding of these aspects, this study is essential to promote person-centered communication about sexual health, addressing the often overlooked needs and concerns of individuals with COPD. Ultimately, the study has the potential to improve sexual health and overall well-being among individuals with COPD, contributing to a more person-centered approach in COPD care.

DETAILED DESCRIPTION:
Objectives The primary objectives of this study are to assess whether impaired sexual health is more prevalent in individuals with COPD compared to those without COPD and to explore its impact on well-being and health-related quality of life. Additionally, the study aims to comprehend the impact of COPD on sexual health by investigating potential associations among selected physical, psychological, and social factors related to sexual health. This understanding is crucial for guiding future studies on identified associations.

The study will examine the following assumptions:

1. Impaired sexual health, characterized by a higher prevalence of sexual dysfunction, dissatisfaction, and distress, is more frequent in individuals with COPD than in a control group (individuals without COPD, matched by age, gender, and relationship status).
2. COPD has a comprehensive impact on both physical, psychological, and social aspects of sexual health. Impaired sexual health is associated with increased loneliness, relationship dissatisfaction, anxiety and/or depression, as well as decreased health-related quality of life and overall well-being.

Method and materials This study adopts a cross-sectional design, utilizing a patient-reported questionnaire to collect data. The participant pool will encompass individuals aged 40 years or older, including those with COPD and a control group without COPD. The control group will be matched to the COPD sample based on age, gender, and relationship status, enhancing the precision of the exploration of COPD-specific challenges. All participants will be invited to complete a public online questionnaire, with all participants providing electronic informed consent before survey completion.

To explore the impact of COPD on sexual health, including COPD-specific factors, and to assess the perceived effect on quality of life, the questionnaire incorporates various validated instruments. Each instrument will measure a specific aspects related to the physical, psychological, or social dimension of sexual health. Sexual dysfunction and sexual health will be assessed using The PROMIS Sexual Function and Satisfaction Measures (Brief Profile), while emotions and concerns related to sexuality will be identified through The Sexual Distress Scale. Relationship dissatisfaction will be assessed using The Couples Satisfaction Index, loneliness through the UCLA Loneliness Scale, and anxiety/depression via the Hospital Anxiety and Depression Scale. Well-being will be evaluated using the EQ-5D-5L. Individuals with COPD will provide additional insights into the impact of COPD on health through the COPD Assessment Test.

Based on a power calculation (two-sided; p<0.05; power=95%) (26), the study's exploratory approach, and the number of variables, a sample size of minimum 200 participants per group is deemed sufficient to identify associations.

Descriptive statistics, including means, standard deviations, and frequencies, will be employed to report the prevalence of sexual health and summarize data related to COPD-specific challenges. Correlation coefficients will be calculated, and multiple regression analyses will be conducted to identify associations between variables, adjusting for potential confounders. STATA will be used for data analysis. The study results will be reported in accordance with the STROBE guidelines (22).

ELIGIBILITY:
Participant inclusion is based upon the reported information provided by the study participants:

Inclusion Criteria:

COPD Population

* Mild to very servere COPD
* ≥40 years old
* Living in Denmark
* Consent to participate the online survey

Control Group:

* Non-COPD, but wit another chronic/longtern disease
* ≥40 years old
* Living in Denmark
* Consent to participate the online survey

Exclusion Criteria:

COPD Population:

* Unwilling to participate and complete the online survey
* Inability to participate and answer the survey questions in Danish due to cognitive impairment, servere illness, or reading or language barriers

Control Group:

* COPD
* Unwilling to participate and complete the online survey
* Inability to participate and answer the survey questions in Danish due to cognitive impairment, servere illness, or reading or language barriers

Ages: 40 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will include individuals aged 40 years or older, encompassing both men and women. The primary focus will be on individuals diagnosed with Chronic Obstructive Pulmonary Disease (COPD), recruited from relevant websites and social media, primarily through the Danish Lung Association platform (www.lungeforeningen.dk). Additionally, a COPD-free control group, controled by age, sex, and relationship status, will serve as a reference group. This comparison group plays a crucial role in identifying COPD-specific challenges. Most non-COPD individuals will be recruited via the 'Aeldresagen.dk' platform. All participants must be capable and willing to complete a public online questionnaire. The study's diverse demographic ensures a comprehensive exploration of COPD-related factors.
Sampling Method: Non-Probability Sample
Enrollment: 521 (Actual)
Dates: Start 2024-02-20 (Actual); Primary Completion 2024-09-19 (Actual); Study Completion 2024-09-19 (Actual)

PRIMARY OUTCOMES:
Sexual health acording to The PROMIS Sex FS BF (vers. 2.0) | Day 1
  The PROMIS® Sexual Function and Satisfaction Measures, version 2.0. Brief Profile (PROMIS SexFS BF v2.0) universally assesses Sexual Function and Satisfaction. A general screener item inquires about sexual activity in the past 30 days. Respondents who have been sexually active answer items covering various domain, e.g. Interest in Sexual Activity, Satisfaction with Sex Life, Orgasm Ability and Pleasure, Erectile Function, Vaginal Discomfort and Lubrication. Most items are gender-nonspecific.
  Higher scores indicate greater Interest, Satisfaction, Orgasm ability, etc. Each domain's summed raw score is converted to T-scores, standardized to the U.S. general population (mean 50, SD 10). A clinically meaningful cutoff is five points below the population mean. (Weinfurt KP et al. J Sex Med. 2015;12:1961-1974.).

SECONDARY OUTCOMES:
Loneliness according to The UCLA Loneliness Scale | Day 1
  Loneliness is assessed by the UCLA Loneliness Scale (revised), a 20 item scale rated on a 4-point Likert scale, ranging from 1 to 4 ('never' to 'always'). The scale covers the frequency of feelings/symptoms related to loneliness and social isolation, assessing three dimensions: emotional, social, and existential loneliness.
  The total sum score ranges from 20 to 80, with higher scores indicating more profound feelings of loneliness.
  (Russell DW. UCLA Loneliness Scale (vers 3). Reliability, validity and factor structure. Journal of Personality Assessment. 1996; 66: 20-40.) (Danish version: Lasgaard M. Reliability and validity of the Danish version of the UCLA Loneliness Scale. Personality and Individual Differences. 2007; 42 (7): 1359-1366.)
Well-being according to EQ-5D-5L Health related quality of life according to the EQ-5D-5L | Day 1
  EuroQoL Five-Dimensional Five-Level Questionnaire (EQ-5D-5L) to assess generic HRQL, by comprising two parts:
  The first part entails five questions covering five domains of life (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) on a 5-item Likert-scale. Participants mark their status from 1 to 5 ('no problems' to 'unable to/extreme problems') for each dimension. Responses are combined to create a five-digit number describing health status (ranging from 11111 to 55555), which is converted to a UI using the EQ-5D-5L value set for Denmark.
  The second part (VAS) assesses the currently experienced health on a vertical VASr between 0 and 100; the latter indicates the best health state imaginable.
  (Jensen CE et al. The Danish EQ-5D-5L Value Set: A Hybrid Model Using cTTO and DCE Data. Appl Health Econ Health Policy. 2021 Jul;19(4):579-591.) (Danish version: Helbredsspørgeskema).
Anxiety and depression according to HADS | Day 1
  The Hospital Anxiety and Depression Scale (HADS) is a 14-item scale consisting of two 7-item subscales assessing anxiety and depression symptoms. Each item is rated on a 4-point Likert scale, ranging from 0 to 3, with higher scores indicating greater levels of anxiety (0-21) and depression (0-21).
  Additionally, a total score for the two components can be summed to provide a composite anxiety-depression score, with a maximum of 42 points. Higher scores indicate more severe symptomatology (Zigmond AS, Snaith RP. The Hospital Anxiety And Depression Scale. Acta Psychiatr Scand 1983; 67: 361-370. DOI: 10.1111/j.1600-0447.1983.tb09716.x) (Danish version: Spørgeskema om angst og depression, til brug på hospital (HADS))
Relationship satisfaction according to The Couples Satisfaction Index | Day 1
  The Couples Satisfaction Index assess relationship satisfaction with 16 items (CSI-16). Comprising 5- and 6-point Likert scale items, respondents are prompted to evaluate their satisfaction across various relationship dimensions.
  The total score, ranging from 0 to 81 (the sum of response point values), indicates the overall level of relationship satisfaction. Higher scores correspond to heightened relationship satisfaction, whereas scores below 51.5 suggest significant relationship dissatisfaction or distress (ibid.).
  (Funk J L; Rogge RD. Testing the ruler with item response theory: Increasing precision of measurement for relationship satisfaction with the Couples Satisfaction Index. Journal of Family Psychology. 2007; 21, 572-583)
  - Trillingsgaard T et al. Relationship Help-Seeking in a Danish Population Sample. J Marital Fam Ther. 2019;45(3):380-394. DOI: 10.1111/jmft.12347 Danish version: "Mål for parforholdstilfredshed".
Sexual distress according to The Sexual Distress Scale | Day 1
  The Sexual Distress Scale - Revised (SDS-R) is utilized to assess sexual distress among both males and females. Sexual distress includes emotions and concerns related to sexuality. The scale comprises 13 items, each using a five-point Likert scale with responses ranging from 0 to 4 ('never' to 'always'). Participants rate the frequency of each feeling/symptom, with higher scores indicating higher sexual distress.
  The total score ranges from 0 to 52, and a cut-off Total score of ≥11 indicates the presence of sexual distress.
  (Santos-Iglesias P et al. A Systematic Review of Sexual Distress Measures. J Sex Med. 2018 May;15(5):625-644. doi: 10.1016/j.jsxm.2018.02.020) (Sood R et al. Association of mindfulness with female sexual dysfunction. Maturitas. 2022 Jul;161:27-32. doi: 10.1016/j.maturitas.2022.02.002.) (Danish version FSDS, 2001)
COPD-impact on health according to CAT | Day 1
  The COPD Assessment Test (CAT) is an 8-item disease-specific questionnaire that assess the impact of COPD on participants' health.
  Each item provides six answer options, with scores ranging from 0 to 5. The total score spans from 0 to 40, with higher values indicating poorer health. A suggested cut-off is CAT <10, reflecting fewer symptoms, and CAT ≥10, indicating more symptoms.
  (Kakavas S, Papanikolaou A, Kompogiorgas S, Stavrinoudakis E, Karayiannis D, Balis E. The Correlation of Sit-to-Stand Tests with COPD Assessment Test and GOLD Staging Classification. COPD. 2020 Dec;17(6):655-661. doi: 10.1080/15412555.2020.1825661.)

CONTACTS AND LOCATIONS:
Overall Officials: Anders L. Ottesen, D.M.Sc., Principal Investigator — Vejle Hospital, Lillebaelt Hospital
Locations (1):
- Vejle Hospital, part of Lillebaelt Hospital, Vejle, Region Syddanmark, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
The plan involves sharing anonymized individual participant data (IPD) from this study to enhance scientific transparency and support further research. Excluding any personally identifiable information such as names, CPR numbers, email addresses, or phone numbers, the shared data will encompass anonymized survey responses, demographic details, and aggregated results at the group level. Efforts will be made to publish the data as supplemental materials in scientific articles, contributing to the broader dissemination of research findings.